CLINICAL TRIAL: NCT00939471
Title: Clinical Evaluation of Confirm the Safety and Efficacy of Balloon Sinuplasty Devices in the Treatment of Pediatric Sinusitis
Brief Title: Safety and Efficacy of Balloon Sinuplasty in Pediatric Sinusitis
Acronym: INTACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integra LifeSciences Corporation (Industry)
Collaborators: Acclarent (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CPR01918
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Relieva™ Balloon Sinuplasty™ System (Other): Balloon Dilation of sinus ostium
  Interventions: Device: Relieva™ Balloon Sinuplasty™ System

INTERVENTIONS:
Device: Relieva™ Balloon Sinuplasty™ System — Balloon dilation will be performed using endoscopic equipment with video documentation capability.
  Other Names: Relieva

SUMMARY:
A non-randomized, multi-center, prospective, clinical study intended to evaluate the safety and efficacy of balloon sinuplasty devices in pediatric patients with longstanding sinusitis following failed medical management.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 2 and < 18 years
2. Both male and female patients eligible
3. Planned surgical intervention (i.e. endoscopic sinus surgery, adenoidectomy, sinus irrigation for obtaining a culture) recommended by PI, consented to by patient's legal guardian)
4. Longstanding sinusitis: >3 mo symptoms OR 6 episodes/yr AND failed 2 courses antibiotics followed by positive CT scan

Exclusion Criteria:

1. Extensive previous sinonasal surgery in target ostia
2. Cystic fibrosis
3. Extensive sinonasal osteoneogenesis
4. Sinonasal tumors or obstructive lesions
5. History of facial trauma that distorts sinus anatomy and precludes access to the sinus ostium
6. Ciliary dysfunction
7. For female patients of childbearing age: the patient is either pregnant or lactating

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2009-07-01 (Actual); Study Completion 2010-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Ramadan, MD, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Balloon Device: Balloon catheter dilation of sinus ostia
Period: Overall Study
Arm/Group | Balloon Device
Started | 44
Completed | 33
Not Completed | 11

BASELINE CHARACTERISTICS:
Arm/Group | Balloon Device
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 44
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.14 (3.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Safety: Device-related Adverse Events During Balloon Dilation Through 12 Months
Description: Number of device-related adverse events from time of procedure through 12 months post-procedure.
Time Frame: 12 months
Measure: Number; unit: number of events
Groups:
- Balloon Sinuplasty Treatment: Balloon catheter dilation of sinus ostia
Arm/Group | Balloon Sinuplasty Treatment
Number analyzed (Participants) | 44
number of events | 0

2. Primary Outcome: Effectiveness: Change in Sinus Symptom Scores (SN-5)
Description: Change in sinus symptoms (mean reduction) for subjects less than 12 years of age evaluated using the SN-5 questionnaire at 52 weeks post-procedure compared to baseline. The maximum possible score for the SN-5 is seven and the minimum is one. A reduction in SN-5 score indicates improvement.
Time Frame: 12 months
Population: Data calculated for matched pairs (subjects with baseline and 12 months follow-up scores).
Measure: Mean (Standard Deviation); unit: change in SN-5 score
Arm/Group | Balloon Sinuplasty Treatment
Number analyzed (Participants) | 23
change in SN-5 score | 2.00 (1.40)

3. Secondary Outcome: Device Success: Ability to Access/Dilate Sinus Ostia
Description: Percentage of sinuses treated which were considered procedure success by the investigator relative to sinuses attempted.
Time Frame: 12 months
Population: intent to treat analysis
Measure: Number; unit: percentage of sinuses successful
Units Other Than Participants: sinuses
Arm/Group | Balloon Sinuplasty Treatment
Number analyzed (Participants) | 44
Number analyzed (sinuses) | 88
percentage of sinuses successful | 90.9

4. Secondary Outcome: Effectiveness: Medication Thru 1 yr
Description: Data was summarized from the Global Patient Assessment Form. Each subject's last observation was used in order to account for any missing data or early termination of subjects. The results indicated represents the proportion of subjects (expressed as a percentage) who reported a decrease in medication usage at the time of their study discontinuation.
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | Balloon Sinuplasty Treatment
Number analyzed (Participants) | 41
percentage of participants | 68.3

5. Secondary Outcome: Effectiveness of Dilation/Measured by Post-op Interventions
Description: Effectiveness of balloon dilation as measured by the need for post-operative interventions other than revision sinus surgery. This endpoint evaluation includes irrigation and debridement. Number of post-operative interventions reported.
Time Frame: 12 months
Measure: Number; unit: number of interventions
Arm/Group | Balloon Sinuplasty Treatment
Number analyzed (Participants) | 44
number of interventions | 0

6. Secondary Outcome: Days Out of School During the 12 Months of Follow-up
Description: Quantitative assessment of days out of school during the 12 months of follow-up.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Balloon Sinuplasty Treatment
Number analyzed (Participants) | 24
days | 5.75 (7.46)

7. Secondary Outcome: Revision Rate
Description: The number of subjects requiring revisions out of 33 subjects treated.
Time Frame: at 1 year
Measure: Number; unit: participants
Arm/Group | Balloon Sinuplasty Treatment
Number analyzed (Participants) | 33
participants | 2

8. Primary Outcome: Effectiveness: Change in Sinus Symptom Scores (SNOT-20)
Description: Change in sinus symptoms (mean reduction) for subjects 12 years of age or greater evaluated using the SNOT-20 questionnaire at 52 weeks post-procedure compared to baseline. The maximum possible score for the SNOT-20 is five and the minimum is zero. A reduction is SNOT-20 score indicates improvement.
Time Frame: 12 months
Population: Data calculated for matched pairs (subjects with baseline and 12 months follow-up scores).
Measure: Mean (Standard Deviation); unit: change in SNOT-20 score
Arm/Group | Balloon Sinuplasty Treatment
Number analyzed (Participants) | 7
change in SNOT-20 score | 0.95 (0.51)

ADVERSE EVENTS:
Arm/Group | Balloon Device
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Scientific Publications Reporting results initiated only by SPONSOR. Sites may not publish single center results before aggregate results. Drafts of abstracts, etc. must be submitted to SPONSOR for review at least sixty (60) days prior to submission for publication. Investigator(s) shall delay submission for up to 90 days to permit patent application filing or shall redact paper to remove language detrimental to SPONSOR's intellectual property interests.